CLINICAL TRIAL: NCT07315412
Title: Comparative Effectiveness of Ginger-Mint and Cinnamon-Flavored Gum in Preventing Nausea and Vomiting Following Pressurized Intraperitoneal Aerosol Chemotherapy
Brief Title: Chewing Gum Flavors to Reduce Postoperative Nausea and Vomiting After PIPAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Collaborators: Istanbul University (Other); Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cansu Mert, Lecturer, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 99.2025fbu
Record Dates: First submitted 2025-12-04; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Nausea and Vomiting (PONV); Peritoneal Metastases From Colorectal Cancer; Intraperitoneal Chemotherapy
Keywords: Chewing gum; ginger; cinnamon; postoperative neusea; vomiting; eras; supportive care
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1:1 ratio to one of three groups (ginger-mint gum, cinnamon gum, or control). Each group receives its assigned intervention in parallel, without crossover.
Masking Description: Because the intervention involves chewing flavored gum, blinding of participants, investigators, and care providers is not feasible. The study will therefore be conducted as an open-label randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ginger-Mint Chewing Gum (Other): Participants chew one piece of ginger-mint flavored, plant-based chewing gum for 15 minutes in the post-anesthesia care unit (PACU).
  Interventions: Other: Ginger-Mint Chewing Gum
- Cinnamon Chewing Gum (Other): Participants chew one piece of cinnamon-flavored, plant-based chewing gum for 15 minutes in the post-anesthesia care unit (PACU).
  Interventions: Other: Cinnamon Chewing Gum
- Standard Postoperative Care (No Intervention): Standard postoperative care, including routine antiemetic prophylaxis, is administered according to the institutional ERAS protocol and is not considered a study intervention.

INTERVENTIONS:
Other: Ginger-Mint Chewing Gum — Participants chew one piece of ginger-mint flavored, plant-based chewing gum (Simply Gum Inc., Brooklyn, NY, USA) for 15 minutes under supervision in the post-anesthesia care unit (PACU) immediately after regaining full consciousness and airway control.
  Arms: Ginger-Mint Chewing Gum
Other: Cinnamon Chewing Gum — Participants chew one piece of cinnamon-flavored, plant-based chewing gum (Simply Gum Inc., Brooklyn, NY, USA) for 15 minutes under supervision in the PACU immediately after regaining full consciousness and airway control.
  Arms: Cinnamon Chewing Gum

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of chewing gum with different natural flavors in reducing postoperative nausea and vomiting (PONV) following Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC). Adult patients undergoing PIPAC will be randomly assigned to one of three groups: (1) ginger-mint flavored gum, (2) cinnamon flavored gum, or (3) control group with standard postoperative care only. Participants in the intervention arms will chew one piece of gum for 15 minutes in the post-anesthesia care unit (PACU). Nausea intensity (Numeric Rating Scale, 0-10) and the presence of vomiting or retching will be assessed at baseline and every 15 minutes for 2 hours.

The study hypothesizes that ginger-mint and cinnamon flavored chewing gums, both plant-based and certified vegan, will be effective, non-pharmacological, and safe methods to reduce nausea and vomiting after PIPAC. This research may contribute to enhanced postoperative comfort and faster recovery by supporting the principles of Enhanced Recovery After Surgery (ERAS).

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) are common and distressing complications in the early postoperative period and remain a significant concern despite routine prophylactic antiemetic use. This problem is particularly relevant in patients undergoing Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC), a minimally invasive but physiologically demanding oncologic procedure associated with increased postoperative discomfort.

Chewing gum has been proposed as a simple, non-pharmacological intervention that may reduce postoperative nausea by stimulating salivation and activating the cephalic-vagal pathway, thereby modulating gastrointestinal function. Previous studies in various surgical populations suggest that gum chewing may contribute to improved postoperative comfort; however, evidence comparing different natural flavors and their potential sensory or acceptability-related effects remains limited.

This study evaluates the comparative effectiveness of ginger-mint-flavored versus cinnamon-flavored chewing gum as an adjunct to standard postoperative care in reducing PONV following PIPAC. By comparing two natural flavors within a controlled clinical setting, the trial aims to explore whether flavor-specific sensory stimulation influences nausea perception and patient experience in the immediate postoperative period.

The findings of this study are expected to contribute to the development of simple, low-cost, and patient-friendly supportive care strategies aligned with Enhanced Recovery After Surgery (ERAS) principles for high-risk surgical populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older undergoing Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC).
* Able to communicate, understand study instructions, and provide written informed consent.
* No known allergy or intolerance to ginger, mint, or cinnamon.
* Able and willing to chew gum for 15 minutes.
* Apfel risk score ≥3 for postoperative nausea and vomiting.

Exclusion Criteria:

* Postoperative complications requiring intensive care or reoperation.
* Need for rescue antiemetic medication within the first 2 postoperative hours.
* History of psychiatric disorder, neurological disease, or cognitive impairment affecting participation.
* Anatomical or functional limitation preventing chewing (e.g., full dentures, jaw restriction, oral surgery).
* Known phenylketonuria or metabolic intolerance to chewing gum ingredients.
* Active chemotherapy, radiotherapy, or immunosuppressive therapy affecting gastrointestinal function.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Nausea Intensity (Numeric Rating Scale, 0-10) | From 0 to 120 minutes postoperatively (measured at baseline, 15, 30, 45, 60, 75, 90, 105, and 120 minutes)
  Nausea intensity will be assessed using the Numeric Rating Scale (NRS, 0-10) where 0 indicates no nausea and 10 indicates the worst possible nausea. The primary endpoint is the change in nausea scores over time (T0-T8). Mean scores and area under the curve (AUC) values will be compared between groups.

SECONDARY OUTCOMES:
Incidence of Vomiting or Retching | 0 to 120 minutes postoperatively
  Presence or absence of vomiting or retching episodes recorded every 15 minutes (T1-T8).
Requirement for Rescue Antiemetic | 0 to 120 minutes postoperatively
  Whether the participant required any rescue antiemetic medication during the 2-hour postoperative observation period (Yes/No).
Patient Acceptability of Chewing Gum | 4 hours postoperatively
  Participants' feedback on taste, comfort, and perceived benefit of the chewing gum, assessed using a brief structured questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Umraniye Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this is a single-center, small-scale interventional study conducted with postoperative patients. The dataset includes sensitive clinical information and cannot be anonymized sufficiently to ensure participant confidentiality. Summary-level results will be made available in publications and upon reasonable request.

REFERENCES:
- [Background] Ge B, Zhao H, Lin R, Wang J, Chen Q, Liu L, Huang Q. Influence of gum-chewing on postoperative bowel activity after laparoscopic surgery for gastric cancer: A randomized controlled trial. Medicine (Baltimore). 2017 Mar;96(13):e6501. doi: 10.1097/MD.0000000000006501. PMID 28353600
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Darvall JN, De Silva AP, von Ungern-Sternberg B, Story DA, Davidson AJ, Allen ML, Tran-Duy A, Schultz-Ferguson C, Ha V, Braat S, Leslie K; CHEWY Trial Group and the ANZCA Clinical Trials Network. Chewing Gum to Treat Postoperative Nausea and Vomiting in Female Patients: A Multicenter Randomized Trial. Anesthesiology. 2025 Mar 1;142(3):454-464. doi: 10.1097/ALN.0000000000005283. Epub 2024 Oct 30. PMID 39476041
- [Background] Mehrabian S, Tirgari B, Beitollahi M, Forouzi MA, Khandani BK. Effect of Cinnamon Essential Oil on the Chemotherapy-Induced Nausea and Vomiting of Cancer Patients. Iran J Nurs Midwifery Res. 2025 Jan 15;30(1):81-86. doi: 10.4103/ijnmr.ijnmr_163_23. eCollection 2025 Jan-Feb. PMID 40052026
- [Background] da Silva RLM, da Silva TTM, Pessoa RL, Sarmento ACA, Medeiros KS, Dantas DV, Dantas RAN. Use of ginger to control nausea and vomiting caused by chemotherapy in patients with cervical cancer undergoing treatment: An experiment. Medicine (Baltimore). 2022 Jun 17;101(24):e29403. doi: 10.1097/MD.0000000000029403. PMID 35713447
- [Background] Efe Erturk N, Tasci S. The Effects of Peppermint Oil on Nausea, Vomiting and Retching in Cancer Patients Undergoing Chemotherapy: An Open Label Quasi-Randomized Controlled Pilot Study. Complement Ther Med. 2021 Jan;56:102587. doi: 10.1016/j.ctim.2020.102587. Epub 2020 Oct 9. PMID 33197662
- [Background] Cetin N, Kose G, Gokbel A. Examining the Effect of Peppermint Oil on Postoperative Nausea After Cervical Surgery. J Neurosci Nurs. 2024 Dec 1;56(6):203-208. doi: 10.1097/JNN.0000000000000790. Epub 2024 Oct 24. PMID 39447066
- [Background] Jaafarpour M, Hatefi M, Najafi F, Khajavikhan J, Khani A. The effect of cinnamon on menstrual bleeding and systemic symptoms with primary dysmenorrhea. Iran Red Crescent Med J. 2015 Apr 22;17(4):e27032. doi: 10.5812/ircmj.17(4)2015.27032. eCollection 2015 Apr. PMID 26023350
- [Background] Zobeiri M, Parvizi F, Shahpiri Z, Heydarpour F, Pourfarzam M, Memarzadeh MR, Rahimi R, Farzaei MH. Evaluation of the Effectiveness of Cinnamon Oil Soft Capsule in Patients with Functional Dyspepsia: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Evid Based Complement Alternat Med. 2021 May 13;2021:6634115. doi: 10.1155/2021/6634115. eCollection 2021. PMID 34093719